CLINICAL TRIAL: NCT05232799
Title: Community Paramedic Hospitalization Reduction and Mitigation Program: Pragmatic Clinical Trial
Brief Title: Care Anywhere With Community Paramedics Program to Reduce Hospitalization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Rozalina G. McCoy, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 21-010816
Record Dates: First submitted 2022-01-27; First posted 2022-02-10 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Acute Illness
Keywords: Community Paramedicine; Acute care; Home care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Care Anywhere with Community Paramedics program (Experimental): Subjects will be discharged from a pre-hospital setting, Emergency Department or the hospital with community paramedic services ordered and overseen by the treating clinical team per current standard of care.
  Interventions: Other: Care Anywhere with Community Paramedics program
- Standard of Care (No Intervention): Subjects will receive continued usual care

INTERVENTIONS:
Other: Care Anywhere with Community Paramedics program — Outpatient management with supportive services provided by the community paramedic team.
  Arms: Care Anywhere with Community Paramedics program

SUMMARY:
The purpose of this research is to compare the effectiveness of the Care Anywhere with Community Paramedics program with usual care in a pragmatic randomized controlled trial. The goal of the Care Anywhere with Community Paramedics program is to prevent or shorten hospitalizations among patients who are being treated in the clinic/ambulatory setting ("prehospital setting"), emergency department, or hospital and are clinically appropriate to be cared for at home with community paramedic services.

DETAILED DESCRIPTION:
This pragmatic randomized controlled trial will randomize, with 1:1 allocation, 240 adults being treated in the pre-hospital setting, emergency department or hospital to either availability of the Care Anywhere with Community Paramedics (CACP) program or to no availability of the CACP program (i.e. usual care). Patients randomized to the CACP program will be able to receive in-home medical care - as ordered by their treating clinicians - from the Mayo Clinic Ambulance Community Paramedic Service. Primary outcome is going to be days alive spent at home without hospitalization (excluding planned admissions), emergency department visits, or skilled nursing facility care.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age ≥ 18 years) patients currently admitted to the ED, hospital or are in a pre-hospital setting but being considered for referral to the ED or hospital in Mayo Clinic Rochester, MN and Barron, WI but do not require hospital-level monitoring or care other than services that could be delivered by CPs in the ambulatory setting.
* Must reside within approximately a 40-mile radius of Rochester, MN or within the service radius of Barron, WI.
* Participants who require assistance with activities of daily living, or who are at increased risk for falls, need to have a caregiver available at home

Exclusion Criteria:

* Referring clinician and the community paramedic service do not believe the patient to be clinically appropriate for outpatient care with the CACP program.
* Inability or unwillingness of individual or legal guardian/representative to give written informed consent.
* Clinical, behavioral, or cognitive instability, determined by the referring clinician or the CACP service.
* Living conditions unsafe for CPs to enter (patient refuses to secure weapons or animals prior to CP's arrival).
* Enrolled in the trial during an earlier hospitalization or ED visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Number of days spent outside the hospital and ED | 30 days
  The number of days spent outside the hospital and ED during the 30 days following enrollment to the trial. (not in the hospital, ED, or nursing home; not counting planned admissions)

SECONDARY OUTCOMES:
Patients with an ED visit hospitalization or death | 30 days
  Proportion of patients with an ED visit, hospitalization, or death within 30-days of the day following randomization
CACP Program patient satisfaction | 30 days
  Percentage of patients who are "extremely likely" or "very likely" to recommend the program
Health related quality of life | 30 days
  EQ-5D survey
Treatment burden | 30 days
  Relevant components of the PETS survey
Community Paramedic satisfaction with the CACP program | 30 days
  CP survey
Referring clinician satisfaction with the CACP program | 30 days
  Clinician Survey

CONTACTS AND LOCATIONS:
Overall Officials: Rozalina McCoy, MD, MS, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Mayo Clinic Health System, Barron, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ridgeway JL, Sundt WJS, Krpata TS, Glasgow A, Smith OA, Lampman MA, Smith-Stellflug JL, Menser TL, Juntunen MB, Liedl CP, Hentz JG, McCoy JJ, McCoy RG. Evaluating adoption and reach in a pragmatic randomized trial of community paramedicine for intermediate acuity patient care. J Clin Transl Sci. 2024 Oct 17;8(1):e199. doi: 10.1017/cts.2024.646. eCollection 2024. PMID 39655042
- [Derived] Ridgeway JL, Gerdes EOW, Dodge A, Liedl CP, Juntunen MB, Sundt WJS, Glasgow A, Lampman MA, Fink AL, Severson SB, Lin G, Sampson RR, Peterson RP, Murley BM, Klassen AB, Luke A, Friedman PA, Buechler TE, Newman JS, McCoy RG. Community paramedic hospital reduction and mitigation program: study protocol for a randomized pragmatic clinical trial. Trials. 2023 Feb 20;24(1):122. doi: 10.1186/s13063-022-07034-w. PMID 36805692
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials